CLINICAL TRIAL: NCT04862052
Title: OPtimal TrEatment for CoroNary Drug Eluting Stent In-Stent Restenosis: Paclitaxel Versus Sirolimus Coated Balloons Versus Everolimus Eluting Stents - the OPEN ISR Study
Brief Title: Optimal Treatment for Coronary Drug Eluting Stent In-stent Restenosis
Acronym: OPEN-ISR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Principal Investigator, Istvan Edes, Associate Professor, Semmelweis University Heart and Vascular Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPEN ISR - 001
Record Dates: First submitted 2021-04-20; First posted 2021-04-27 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Coronary Stent Restenosis
Keywords: drug eluting stent; restenosis; drug coated balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Xience chromium-cobalt everolimus eluting stent (Active Comparator): The Xience chromium-cobalt everolimus eluting stent will be evaluated in prior implanted coronary drug eluting stent restenosis.
  Interventions: Procedure: Intravascular management of prior implanted coronary drug eluting stent restenosis
- Emperor paclitaxel coated balloon (Experimental): The Emperor paclitaxel coated balloon will be evaluated in prior implanted coronary drug eluting stent restenosis.
  Interventions: Procedure: Intravascular management of prior implanted coronary drug eluting stent restenosis
- Magic Touch sirolimus coated balloon (Experimental): The Magic Touch sirolimus coated balloon will be evaluated in prior implanted coronary drug eluting stent restenosis.
  Interventions: Procedure: Intravascular management of prior implanted coronary drug eluting stent restenosis

INTERVENTIONS:
Procedure: Intravascular management of prior implanted coronary drug eluting stent restenosis — Intravascular devices will be assessed for the management of prior implanted drug eluting stent restenosis management.

SUMMARY:
The aim of this open label, randomized study is to compare the safety and efficacy of three different methods to handle coronary drug eluting stent (DES) in-stent restenosis (ISR).

These are the:

* Magic Touch - sirolimus coated balloon
* Emperor - paclitaxel and dextran coated balloon
* Xience - chromium-cobalt everolimus eluting stent

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for intervention of drug eluting stent restenosis
* Restenosis suitable for all three treatment arms as per 'instructions for use' of the devices
* Optional enrollment in the optical coherence tomography sub-study (10-20% of patients)

Exclusion Criteria:

* Patients undergoing coronary angiography after sudden cardiac death
* Pregnant or nursing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of new onset target vessel myocardial infarction | 6 months
  New onset myocardial infarction that affects the target vessel treated with either study device
Occurrence of target vessel revascularization of failure | 6 months
  The need for further revascularization affecting the target vessel treated with either study device, or the failure of the vessel treated by either study device.
Occurrence of target lesion revascularization | 6 months
  The need for further revascularization of the target lesion after treatment with either study device.

SECONDARY OUTCOMES:
Percentage late lumen loss | 6 months
  Late lumen loss measured via qualitative coronary angiography in treated segment(s)
Percentage intraluminal gain after treatment | index procedure
  Intraluminal gain after assigned treatment measured via optical coherence tomography
Square millimetre intraluminal gain after treatment | index procedure
  Intraluminal gain after assigned treatment measured via optical coherence tomography
Percentage intraluminal gain after treatment | 6 months
  Intraluminal gain after assigned treatment measured via optical coherence tomography
Square millimeter intraluminal gain after treatment | 6 months
  Intraluminal gain after assigned treatment measured via optical coherence tomography
Endothelium coverage in micrometers | 6 months
  Mean endothelium thickness of stent struts in micrometres measured via optical coherence tomography
Late lumen loss in square millimetres | 6 months
  Late lumen loss in square millimetres measured via optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: István F Édes, MD PhD, Principal Investigator — Semmelweis University Heart and Vascular Center
Locations (2):
- Hungary (2):
  - Semmelweis University Heart and Vascular Center, Budapest, Budapest
  - University of Szeged, Department of Invasive Cardiology, Szeged, Csongád-Csanád

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kulyassa P, Nemeth BT, Ehrenberger R, Ruzsa Z, Szuk T, Fehervari P, Engh MA, Becker D, Merkely B, Edes IF. The Design and Feasibility of the: Radial Artery Puncture Hemostasis Evaluation - RAPHE Study, a Prospective, Randomized, Multicenter Clinical Trial. Front Cardiovasc Med. 2022 May 27;9:881266. doi: 10.3389/fcvm.2022.881266. eCollection 2022. PMID 35694680
- [Derived] Kulyassa PM, Nemeth BT, Hizoh I, Janko LK, Ruzsa Z, Jambrik Z, Balazs BB, Becker D, Merkely B, Edes IF. The Design and Feasibility of Optimal Treatment for Coronary Drug-Eluting Stent In-Stent Restenosis (OPEN-ISR)-A Prospective, Randomised, Multicentre Clinical Trial. J Pers Med. 2025 Feb 2;15(2):60. doi: 10.3390/jpm15020060. PMID 39997337
- See also: Link to design and feasibility manuscript — https://www.frontiersin.org/articles/10.3389/fcvm.2022.881266/full